CLINICAL TRIAL: NCT04923659
Title: Pharmacological Mechanisms of Low-intensity Focused Ultrasound for Motor Cortex Neuroplasticity
Acronym: LIFUS-Pharma
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Robert Chen, Senior Neurologist and Scientist, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: YS609220
Record Dates: First submitted 2021-05-25; First posted 2021-06-11 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Low Intensity Focussed Ultrasound
MeSH Terms: interventions — Carbamazepine; Lorazepam; Dextromethorphan; Acetylcysteine; Nimodipine; Sugars

STUDY DESIGN:
Masking Description: Healthy Controls 18-80 years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- LIFUS (Experimental): Low Intensity Focussed ultrasound.
  Interventions: Drug: Carbamazepine; Drug: Lorazepam; Drug: Dextromethorphan; Drug: Nimodipine; Drug: Placebo

INTERVENTIONS:
Drug: Carbamazepine — 600 mg reconstituted as one table. Administered once
  Other Names: Tegretol
Drug: Lorazepam — 2.5 mg mg reconstituted as one table. Administered once
  Other Names: Ativan
Drug: Dextromethorphan — 150 mgmg reconstituted as one table. Administered once
  Other Names: Robitussin
Drug: Nimodipine — 30 mg reconstituted as one table. Administered once
  Other Names: Nimotop
Drug: Placebo — Administered once
  Other Names: Sugar

SUMMARY:
Low-intensity focused ultrasound (LIFUS) has been shown to be an effective and safe non-invasive brain stimulation technique, capable of reaching greater brain depth and a greater spatial resolution than other brain stimulation tools. Its use as a potential clinical tool for treatment of neurological disorders is reliant on an understanding of its mechanisms of action. Although it has been shown to induce immediate (online) and prolonged (offline) changes in plasticity in the motor cortex, researchers have not studied its effects on neurotransmitter receptors and ion channels responsible for neuronal signaling in humans. The purpose of this study is to explore the effects of online and offline LIFUS stimulation in tandem with administration of various brain-active drugs, to elucidate the effects of this technique on specific cortical receptors and channels. 20 healthy, screened subjects will be recruited to participate in 5 sessions in-lab. Each session will represent the double-blinded administration of four known and studied pharmacological agents known to safely induce changes in the motor cortex, as well as a placebo. Investigators will use carbamazepine (sodium channel blocker), lorazepam (GABAA positive allosteric modulator), nimodipine (calcium channel blocker), and dextromethorphan (glutamate N-Methyl-D-aspartate receptor antagonist). Single- and paired-pulse transcranial magnetic stimulation (TMS) measures will be recorded for online LIFUS before and after drug intervention, and induction of offline LIFUS during placebo will be compared with its induction following the various drug interventions. Investigators predict that due to the differential effects of online and offline LIFUS on motor parameters, the mechanisms in which it alters the receptors and channels of interest will also be differentially modulated.

DETAILED DESCRIPTION:
In the current study investigators aim to describe how common neurotransmitter receptors and ion channels in the brain, particularly the motor cortex, are dynamically involved in the mechanisms generated by LIFUS. By selectively modulating the activity of these receptors and channels with previously studied and known drugs, it can be empirically determined how common components of signal propagation and prolonged neuroplasticity are being affected by the sonication waves induced by LIFUS. This will be done through baseline recording of FUS-induced neuroplasticity, and then compared within-subject to FUS-induced neuroplasticity after administration of pharmacological agents of interest. Random double-blinded administration of four drugs and a placebo will ensure that results are accurate and reduce any effects of expectation. Its predicted that online FUS will lead to a reduction in motor excitation and an increase in intracortical inhibition, and offline FUS will lead to an increase in motor excitation, an increase in intracortical facilitation, and a reduction in intracortical inhibition. Its predicted that drugs of interest to similarly replicate previous work; that is, carbamazepine, lorazepam, dextromethorphan, and nimodipine will all reduce cortical excitation and increase intracortical inhibition compared to placebo. Its predicted that carbamazepine, lorazepam, nimodipine and dextromethorphan will all further reduce motor excitation in conjunction with online FUS in an additive manner, compared to placebo. Its predicted that carbamazepine will have no effect on the prolonged effects of offline FUS on the motor cortex, but that lorazepam, nimodipine, and dextromethorphan will all interfere with the offline effects of FUS on motor cortex, compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed healthy subjects between the ages of 18-65 will be included for recruitment.

Exclusion Criteria:

* Diagnosed with any gait or postural disorders
* Major neurological disease or disorder
* Major musculoskeletal or nerve disorder, or disorder of hands, wrists and upper limbs
* History of stroke or seizure
* Diagnosed with dementia
* Diagnosed with myasthenia gravis or acute narrow angle glaucoma
* Has intracranial implant(s) or device(s)
* Has an implanted cardiac pacemaker or implantable cardioverter-defibrillator (ICD)
* Presence of metal implanted in body that is contraindicated in TMS
* Caffeine or chocolate consumption 1-2 hours before study sessions
* Consumption of grapefruit juice 24 hours before study sessions
* Alcohol consumption 24 hours before study sessions
* Pregnancy*
* Major depression/psychiatric disorder that in the opinion of the Investigator will affect patient's understanding of study procedures and willingness to abide by all procedures during the course of the study
* Regular usage of CNS active drugs or calcium channel blockers during or up to 2 weeks before participating in the study**
* Is on antipsychotics, marijuana, or other recreational drugs (including tobacco) that affect the nervous system
* Major cardiac, hematopoietic, liver, or kidney disease or infection
* Treated hypertension
* Hypersensitivity to benzodiazepines
* Hypersensitivity to calcium channel blockers
* Hypersensitivity to antitussives
* Hypersensitivity to anticonvulsants
* Regular usage of androgens, antibiotics, antifungals, antivirals, cardiovascular/gastrointestinal drugs, muscle relaxants, and platelet aggregation inhibitors during or up to 2 weeks before participating in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2022-07-10 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Motor Evoked Potential | 2 years
  1 mV peak-to-peak MEP (motor evoked potential), defined as the average TMS stimulation intensity required to elicit a 1-mV EMG response in the right hand muscle. We will compare the intensities required to elicit this response within all of our pharmacological and FUS interventions, compared to our sham/placebo FUS intervention.
Resting Motor Threshold | 2 years
  • The resting motor threshold (RMT) is defined as the minimum stimulus intensity that elicits an MEP greater than or equal to 50 microvolts in at least 5 out of 10 trials in the relaxed right FDI. We will compare the RMT required to elicit this response within all of our pharmacological and FUS interventions, compared to our sham/placebo FUS intervention.
Recruitment Curve | 2 years
  • The MEP recruitment curve is a dose-response curve for assessing the effects of TMS stimulation intensity on recorded MEP. TMS stimulation begin at sub-RMT levels (80-90%) and is increased in increments of 10%. During this, MEP response is recorded from the right FDI, and a graph may then be created by fitting data-points into a sigmoidal curve. Recruitment curves will be compared in-between sham and real FUS, and in-between our various pharmacological interventions to observe changes in cortical neuron activation.
Short Interval Intracortical Inhibition | 2 years
  • Short Interval Intracortical Inhibition (SICI) will be obtained on a relaxed right FDI muscle using paired-pulse TMS. SICI involves a subthreshold conditioning stimulus (CS) at 80% of RMT followed by a suprathreshold test stimulus (TS) at an intensity able to evoke an average MEP of ~1mV, at an interstimulus interval of 2ms. The magnitude of SICI will be indexed by the ratio of the mean conditioned MEP amplitude over the mean unconditioned MEP amplitude. A ratio less than 1 indicates greater inhibition and less facilitation.
Intracortical Facilitation | 2 years
  • Intracortical Facilitation (ICF) will be obtained on a relaxed right FDI muscle using paired-pulse TMS. ICF involves a subthreshold conditioning stimulus (CS) at 80% of RMT followed by a suprathreshold test stimulus (TS) at an intensity able to evoke an average MEP of ~1mV, at an interstimulus interval of 10ms. The magnitude of ICF will be indexed by the ratio of the mean conditioned MEP amplitude over the mean unconditioned MEP amplitude. A ratio greater than 1 indicates greater facilitation and less inhibition.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Chen, MBBS, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No